CLINICAL TRIAL: NCT01363427
Title: Retrospective Data Analysis of Newly Diagnosed Crohn's Disease Patients in Gastroenterological Surgeries
Brief Title: Retrospective Data Analysis in Crohn's Disease
Acronym: Crohn 2
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Other Study IDs: FE 999907 (Pentasa)
Record Dates: First submitted 2011-05-30; First posted 2011-06-01 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Crohn's disease: Patients with initially diagnosed Crohn's disease

SUMMARY:
The purpose of this study is to identify prognostic parameters about efficacy of Mesalazine in recently diagnosed patients with Morbus Crohn by retrospective data collection.

ELIGIBILITY:
Inclusion Criteria:

* therapeutic need according to SPC
* written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Private practices
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2007-03; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Response to Mesalazine: measured by time to step up therapy | 12 to 48 months

SECONDARY OUTCOMES:
Identification and characterisation of the responding sub-population | 12 to 48 months
  measured by: (a) Age at diagnosis, (b) Proportion of patients with minor endoscopic lesions, (c) Lack of severe mucosal lesions (Adapted Rutgeerts Score < 2)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (16):
- Germany (16):
  - Investigational Site, Ehrenfelsstraße 47, Berlin
  - Investigational Site, Möllendorfstraße 111, Berlin
  - Investigational Site, Graseggerstraße 105, Cologne
  - Investigational Site, Münchner Straße 64, Dachau
  - Investigational Site, Karlsbader Straße 7, Dinkelsbühl
  - Investigational Site, Heiligengrabstraße 16, Hof
  - Investigational Site, Am Tiefen Weg 2, Karlstadt am Main
  - Investigational Site, Erdbeerfeld 8, Kiel-Altenholz
  - Investigational Site, Hohenfelder Straße 20, Koblenz
  - Investigational Site, Funkenburgstraße 19, Leipzig
  - Investigational Site, Franz-Kail-Straße 2, Leverkusen
  - Investigational Site, Bahnhofplatz 2, Mainz
  - Investigational Site, Uferstraße 3, Minden
  - Investigational Site, Hammer Straße 95, Münster
  - Investigational Site, Weiltinger Str. 11, Nuremberg
  - Investigational Site, Marktplatz 23, Rottenburg